CLINICAL TRIAL: NCT02855697
Title: Single Arm Feasibility of Multi-maintenance Olaparib After Disease Recurrence in Participants With Platinum Sensitive BRCAm High Grade Serous Ovarian Cancer
Brief Title: Multi-maintenance Olaparib After Disease Recurrence in Participants With Platinum Sensitive BRCAm High Grade Serous Ovarian Cancer
Acronym: MOLTO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Clinical Trials Unit, Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15_DOG01_142
Record Dates: First submitted 2016-07-25; First posted 2016-08-04 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; cediranib; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib +/- cediranib (Experimental): Patients are administered two courses of maintenance olaparib following chemotherapy. It is possible for patients to take cediranib during the second course of olaparib if recommended as per the protocol.
  Interventions: Drug: Olaparib; Drug: Cediranib; Drug: Platinum-based Chemotherapy

INTERVENTIONS:
Drug: Olaparib — 300 mg taken twice daily, equivalent to a total daily dose of 600 mg
  Other Names: Lynparza; AZD2281; KU-0059436
Drug: Cediranib — 20mg dose of cediranib was selected for this study
  Other Names: AZD2171
Drug: Platinum-based Chemotherapy — 1 or 2 two courses of platinum-based chemotherapy administered depending on trial entry point.

SUMMARY:
PARP inhibitors, such as olaparib, significantly improve progression free survival (PFS) in participants with recurrent, platinum-sensitive high-grade serous/endometrioid ovarian cancer (HGS/EOC), who harbour a germline mutation in BRCA 1 or 2 genes. Despite some of the most impressive hazard ratios seen in ovarian oncology, such improvements in PFS have not translated into improved overall survival (OS) advantage potentially because maintenance poly ADP ribose polymerase inhibitors (PARPi) are only being administered during a single remission. Here the investigators will test the feasibility of administering a second course of olaparib in participants who have recurrent platinum-sensitive HGS/EOC.

DETAILED DESCRIPTION:
Epithelial ovarian cancer presents in most participants at an advanced stage when curative surgery is not possible because of extensive pelvic, abdominal or distant metastases. Immediate or delayed surgery combined with platinum-based chemotherapy are the standards of care but even with complete surgical cytoreductive techniques and the prescription of combination platinum-based chemotherapy, the 5 year survival rate remains approximately 35%.

Approximately 50% of ovarian cancers harbour defects in HR. Defects in the pathway can arise as a result of genomic or epigenetic events in any one of up to 33 genes.

Phase I and II clinical trials with the PARPi, olaparib, have shown promising results in BRCA mutated (BRCAm) recurrent EOC and in a proportion of HGSOC participants with wild type germline BRCA (BRCA wt). Additionally the favourable toxicity profile of olaparib has prompted the long-term use of PARPi as a maintenance strategy. The results of a randomized placebo-controlled phase II clinical trial of olaparib maintenance therapy showed an improvement in progression free survival (PFS) and time to progression in participants with recurrent platinum-sensitive HGSOC6. Recent data have confirmed that the increase in median PFS is most marked in BRCAm participants who received olaparib as maintenance treatment compared with the BRCAm participants who received placebo treatment (11.2 vs 4.3 months respectively; HR, 0.18; 95% CI, 0.11-0.31; p<0.00001). These studies were performed with the original capsule formulation of olaparib at a dose of 400mg bd.

Rationale for this study The improvement in PFS with maintenance olaparib in participants with germline BRCA-mutation (g-BRCAm), although particularly striking, has not translated into improved overall survival, presumably because subsequent salvage therapy obscures this effect. Emerging data indicate that a significant proportion of BRCAm HGSOC participants retain sensitivity to platinum agents or other chemotherapies following progression on olaparib. Thus it is appropriate to offer further platinum-containing therapy to participants whose disease progresses more than 6 months after previous platinum therapy. In those whose disease benefits from further platinum chemotherapy, a further course of olaparib might consolidate the gains from the first course of olaparib, improving PFS to the point that OS is increased as well. However, to date no trial has tested the feasibility of successive treatments with 2 or more courses of maintenance olaparib and this issue will be addressed here, in participant who harbour a germline BRCA defect and whose disease has recurred and which is at least stabilised by subsequent platinum-based chemotherapy.

Functional testing remains the gold standard test for HR status and has greater predictive accuracy than non-functional tests. The Rad51 functional assay involves the recognition of completion of HR by the formation of Rad51 foci in viable cells that have undergone DNA damage, recognised by γH2AX focus formation. The assay is robust and reproducible but requires viable cells derived from either participant ascites or solid tumour deposits.

ELIGIBILITY:
Inclusion Criteria:

1. Progressive, measureable high grade serous or endometrioid ovarian cancer, fallopian tube or primary peritoneal cancer

   * Participants who have not been treated with PARP inhibitor previously will be treated with two maintenance courses of olaparib.
   * Participants, who have received one course of maintenance olaparib before entry to the trial, will only receive one further course of treatment.
2. Aged 18 or over
3. Measureable disease by RECIST 1.1
4. ECOG performance status 0-2 and life expectancy of over 12 weeks
5. Adequate haematological function: Hb ≥ 10.0 g/l, Neutrophils ≥ 1.5 x 109/l, Platelets ≥ 100 x 109/l; coagulation: INR <1.4 (unless therapeutically anti-coagulated) and/or APPT ratio <1.4
6. Adequate liver function: bilirubin ≤1.5 x ULN, Transaminases (ALT and AST) ≤2.5x ULN unless liver metastases are present in which case they must be ≤ 5x ULN
7. Adequate renal function defined as GFR ≥ 51ml/min
8. Written, informed consent that includes genetic research on tissue derived from biopsies.
9. Pathogenic germline BRCA-1 or -2 gene mutation
10. Ability to swallow oral medication (tablets).

Exclusion Criteria:

1. Concurrent medical illness that would impact on compliance with the protocol including MDS/ AML
2. Uncontrolled brain metastases or seizures. A scan to confirm the absence of brain metastases is not required.
3. Known positivity for Hep B, Hep C or HIV.
4. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
5. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
6. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
7. Another cancer, which has been active within the previous 5 years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin and no evidence of recurrence of other malignancy.
8. Female participants who are able to become pregnant (or are already pregnant or lactating) unless the following apply: Those who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for one month afterwards are considered eligible. Alternatively if the participant can abstain from sexual intercourse for the same interval, then they are eligible to participate.
9. Participants who are planning to receive maintenance bevacizumab.
10. Participants will be excluded if the side effects of previous treatments have not resolved to grade I or less, with the exception of alopecia or grade 2 neurotoxicity that is considered related to cytotoxic chemotherapy.
11. Radiotherapy, surgery or tumour embolization within 28 days before the cycle 1 day 1 of the platinum-containing chemotherapy.
12. Additional concurrent anti-cancer therapy.
13. Causes of malabsorption e.g. uncontrolled diarrhoea or poorly controlled stoma is not permitted.
14. Participants who have contra-indications to VEGF inhibitors will not be eligible to receive cediranib (second treatment). These contra-indications include concurrent or past history of malignant fistula, uncontrolled hypertension, recent arterial thrombosis (cerebrovascular accident or myocardial infarction) within the past 6 months, participants who are at risk of bowel perforation, proteinuria greater than 2g/24 hours or a past history of VEGF inhibitor-associated reversible posterior leukoencephalopathy.
15. Any participant that is participating in another interventional clinical trial within 30 days or 5-lives prior to signing of consent. Participation in an observational trial would be acceptable.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of administering a second course of maintenance olaparib for more than 6 months (26 weeks) to participants with recurrent platinum-sensitive HGS/EOC who have been previously treated with olaparib. | 6 months after the last patient has started the second course of olaparib
  The proportion of participants who remain on olaparib for more than 6 months (26 weeks) in the second course of maintenance olaparib.

SECONDARY OUTCOMES:
Impact of multi-maintenance olaparib treatment on time to first subsequent therapy (TFST) in participants with platinum sensitive recurrent BRCAm HGS/EOC. | 6 months after the last event
  Secondary endpoints will include time to first subsequent chemotherapy (TFST), which is defined as the interval from the last day of the last cycle of a prior regimen of chemotherapy to the first day of the first cycle of the subsequent regimen for each course of chemotherapy, following the first course of olaparib.
Impact of multi-maintenance olaparib treatment on time to second subsequent therapy (TSST) in participants with platinum sensitive recurrent BRCAm HGS/EOC. | 6 months after the last event
  Secondary endpoints will include time to second subsequent chemotherapy (TSST), which is defined as the interval from the last day of the last cycle of a prior regimen of chemotherapy to the first day of the first cycle of the subsequent regimen for each course of chemotherapy, following the second course of olaparib.
Progression-free survival (PFS) for each course of chemotherapy followed by olaparib | 6 months after the last event
  Secondary endpoints will include PFS for each course of chemotherapy, which is followed by olaparib.

OTHER OUTCOMES:
To evaluate the feasibility of obtaining fresh tissue biopsies before each course of platinum chemotherapy, where the intention is to maintain platinum-induced clinical benefit with olaparib. | 6 months after the last patient starts the second course of olaparib.
  The proportion of biopsies received from the total number of patients who begin each course of platinum-based chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, MD, Prof., Study Chair — The Christie National Health Service (NHS) Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom